CLINICAL TRIAL: NCT00193128
Title: A Phase I/II Trial of Preoperative Oxaliplatin, Docetaxel, and Capecitabine With Concurrent Radiation Therapy in Localized Carcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Preoperative Therapy With Oxaliplatin/Docetaxel/Capecitabine and Radiation in Resectable Esophagus Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Sanofi-Synthelabo (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 57
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Esophagus Cancer
Keywords: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; Docetaxel; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Oxaliplatin 40 mg/m2 intravenously (IV) over 2 hours and docetaxel 20 mg/m2 IV over 30 minutes on days 1, 8, 15, 22, and 29. Radiation therapy began concurrently with day 1 of chemotherapy at a dose of 1.8 Gy/d Monday through Friday to a total of 45 Gy (25 fractions).
  Patients were to have esophageal resection after completion of preoperative therapy during weeks 9 to 12 and after all treatment-related side effects were resolved.
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Radiation: Radiation therapy
- Cohort 2 (Experimental): Oxaliplatin 40 mg/m2 intravenously (IV) over 2 hours and docetaxel 20 mg/m2 IV over 30 minutes on days 1, 8, 15, 22, and 29. Capecitabine was administered 1000 mg/m2 orally twice daily on days 1 to 7, 15 to 21, and 29 to 35. Radiation therapy began concurrently with day 1 of chemotherapy at a dose of 1.8 Gy/d Monday through Friday to a total of 45 Gy (25 fractions).
  Patients were to have esophageal resection after completion of preoperative therapy during weeks 9 to 12 and after all treatment-related side effects were resolved.
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Drug: Capecitabine; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Oxaliplatin — 40 mg/m2 IV over 2 hours on days 1, 8, 15, 22, and 29 in both treatment cohorts
  Other Names: Eloxatin
Drug: Docetaxel — 20 mg/m2 IV over 30 minutes was administered on days 1, 8, 15, 22, and 29 in both cohorts
  Other Names: Taxotere
Drug: Capecitabine — In Cohort 2, capecitabine was administered 1000 mg/m2 orally twice daily on days 1 to 7, 15 to 21, and 29 to 35.
  Other Names: Xeloda
  Arms: Cohort 2
Radiation: Radiation therapy — In both cohorts, radiation therapy began concurrently with day 1 of chemotherapy at a dose of 1.8 Gy/d Monday through Friday to a total of 45 Gy (25 fractions).
  Other Names: RT

SUMMARY:
In this phase I/II trial, we will evaluate a novel combination of chemotherapy, used concurrently with radiation therapy, in the preoperative therapy of locoregional carcinoma of the esophagus and gastroesophageal junction. In the brief phase I portion of this trial, we will determine whether 2 drugs (docetaxel/oxaliplatin) or 3 drugs (docetaxel/oxaliplatin/capecitabine) can be used concurrently with radiation therapy. If the 3-drug regimen is tolerated, the phase II portion will proceed with this regimen. If the 3-drug combination is considered too toxic, the phase II study will proceed with docetaxel/oxaliplatin in combination with radiation therapy.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

Oxaliplatin + Docetaxel + Capecitabine + Radiation therapy

If the three-drug chemotherapy regimen, with radiation therapy, is tolerable, this regimen will be taken forward into the phase II portion of the trial. If the three-drug regimen is too toxic, the phase II portion will proceed with the two-drug regimen Oxaliplatin + Docetaxel + Radiation therapy

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Adenocarcinoma or squamous cell carcinoma of the esophagus or G/E junction.
* Must be surgical candidates
* No previous treatment for esophageal cancer
* Must have measurable or evaluable disease
* Able to perform activities of daily living with minimal to no assistance
* Adequate bone marrow, liver and kidney function
* Provide written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Tumor location in the proximal esophagus
* Metastatic disease or locally advanced cancer
* Moderate to severe peripheral neuropathy
* Serious pre-existing medical illnesses
* Significant heart disease
* Treated for an invasive cancer within the previous 5 years
* Women who are pregnant or breast-feeding
* Age < 18 years

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-04; Primary Completion 2008-02 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Tower Oncology, Beverly Hills, California
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Atlanta Cancer Care, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Greco FA, Meluch AA, Lane CM, Farley C, Gray JR, Clark BL, Burris HA 3rd, Hainsworth JD. Phase I/II trial of preoperative oxaliplatin, docetaxel, and capecitabine with concurrent radiation therapy in localized carcinoma of the esophagus or gastroesophageal junction. J Clin Oncol. 2010 May 1;28(13):2213-9. doi: 10.1200/JCO.2009.24.8773. Epub 2010 Mar 29. PMID 20351330
- See also: Published article in the Journal of Clinical Oncology — http://jco.ascopubs.org/cgi/reprint/28/13/2213

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaliplatin/Docetaxel/Radiation (Cohort 1): oxaliplatin, docetaxel and radiation therapy
  Ten patients were enrolled on the phase I cohort 1 portion of the trial. The combination was tolerated and phase I cohort 2 subsequently began.
- Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2): Oxaliplatin, docetaxel, capecitabine, and radiation therapy.
  Ten patients were enrolled in phase I cohort 2; an additional 39 patients were subsequently enrolled in the phase II portion and treated with the phase I cohort 2 regimen. Data from all 49 patients receiving the cohort 2 regimen was analyzed and reported.
Period: Overall Study
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2)
Started | 10 | 49
Completed | 10 | 39
Not Completed | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2) | Total
Number analyzed (Participants) | 10 | 49 | 59
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 77] | 63 [42 to 81] | 61 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 8 | 41 | 49
Region of Enrollment [Number; unit: participants]
  United States | 10 | 49 | 59

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (PCRR), the Percentage of Patients Who Have No Evidence of Cancer in Their Surgical Specimen Following Surgery
Description: The absence of any residual tumor cells in a histologic evaluation of a tumor specimen following surgery is defined as a complete pathologic response
Time Frame: 18 months
Population: Analysis was conducted on the 49 patients in Cohort 2 who received triplet chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Oxaliplatin/Docetaxel/Radiation (Cohort 1): Oxaliplatin, docetaxel, and radiation therapy.
  Ten patients were enrolled on the phase I cohort 1 portion of the trial. The combination was tolerated and phase I cohort 2 subsequently began.
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2)
Number analyzed (Participants) | 0 | 49
Participants |  | 24

2. Secondary Outcome: Disease-Free Survival (DFS)
Description: Defined as the interval between the start date of treatment and the date of occurrence of progressive disease or death from any cause.
Time Frame: 18 months
Population: Analysis was conducted on the 49 patients in Cohort 2 who received triplet chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2)
Number analyzed (Participants) | 0 | 49
months |  | 16.3 [4.5 to 31.5]

3. Secondary Outcome: Overall Survival (OS)
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until death.
Time Frame: 36 months
Population: Analysis was conducted on the 49 patients in Cohort 2 who received triplet chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Oxaliplatin/Docetaxel/Radiation (Cohort 1): oxaliplatin, docetaxel and radiation therapy
  Oxaliplatin, docetaxel, and radiation therapy.
  Ten patients were enrolled on the phase I cohort 1 portion of the trial. The combination was tolerated and phase I cohort 2 subsequently began
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2)
Number analyzed (Participants) | 0 | 49
months |  | 24.1 [11.4 to 36]

ADVERSE EVENTS:
Arm/Group | Oxaliplatin/Docetaxel/Radiation (Cohort 1) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 2/10 | 33/49
Other Adverse Events (participants affected / at risk) | 10/10 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin/Docetaxel/Radiation (Cohort 1) (N=10) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2) (N=49)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 4 (5)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Infection - Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Respiratary - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pneumoperitoneum
Dehydration (Gastrointestinal disorders) | 0 (0) | 6 (6)
Perforation, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fistula, GI (Gastrointestinal disorders) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain - Abdomen (General disorders) | 0 (0) | 1 (1)
Stricture, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GI - Other (Gastrointestinal disorders) | 0 (0) | 1 (2) — Hematemesis
Pain - Back (General disorders) | 0 (0) | 1 (1)
CNS Ischemia (Nervous system disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Paraesophageal hernia
Infection - Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin/Docetaxel/Radiation (Cohort 1) (N=10) | Oxaliplatin/Docetaxel/Capecitabine/Radiation (Cohort 2) (N=49)
Hemoglobin (Blood and lymphatic system disorders) | 3 (6) | 19 (51)
Anorexia (Gastrointestinal disorders) | 5 (12) | 23 (101)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (6)
Pain - joint (General disorders) | 1 (1) | 0 (0)
Cold intolerance (General disorders) | 2 (6) | 3 (9)
Constipation (Gastrointestinal disorders) | 2 (3) | 16 (45)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 23 (63)
Pain - abdomen (General disorders) | 1 (2) | 0 (0)
Pain - chest (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 3 (8)
Dysphagia (Gastrointestinal disorders) | 3 (15) | 19 (76)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 3 (14) | 25 (92)
Fistula - esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (38) | 36 (171)
Fever (General disorders) | 1 (1) | 13 (26)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (5) | 6 (10)
Hypotension (Cardiac disorders) | 2 (5) | 4 (17)
Insomnia (General disorders) | 1 (5) | 9 (22)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 1 (2) | 15 (32)
Nausea (Gastrointestinal disorders) | 7 (22) | 35 (112)
Neuropathy (Nervous system disorders) | 3 (18) | 5 (9)
Infection - pneumonia (Infections and infestations) | 1 (1) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (18)
Infection - sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 3 (6) | 19 (47)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 20 (36)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (14)
Dehydration (Gastrointestinal disorders) | 0 (0) | 19 (42)
Edema NOS (Blood and lymphatic system disorders) | 0 (0) | 3 (9)
Gastroesophageal reflux disorder (Gastrointestinal disorders) | 0 (0) | 3 (5)
Heartburn (Gastrointestinal disorders) | 0 (0) | 3 (8)
Infection NOS (Infections and infestations) | 0 (0) | 9 (18)
Mucositis (Gastrointestinal disorders) | 0 (0) | 5 (9)
Pain NOS (General disorders) | 0 (0) | 3 (7)
Pain - throat (General disorders) | 0 (0) | 7 (34)
Weight loss (General disorders) | 0 (0) | 5 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.